CLINICAL TRIAL: NCT03809221
Title: The Effectiveness and Safety of the Early Follicular Phase Prolonged Down-regulation Protocol for Controlled Ovarian Hyperstimulation: a Randomized, Paralleled, Controlled, Multicenter Trial
Brief Title: The Effectiveness and Safety of the Prolonged Down-regulation Protocol for Controlled Ovarian Hyperstimulation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Peking University People's Hospital (Other)
Collaborators: West China Hospital (Other); Peking University First Hospital (Other); The First Affiliated Hospital of Zhengzhou University (Other); Henan Provincial People's Hospital (Other); The Second Hospital of Hebei Medical University (Other); First Affiliated Hospital of Wenzhou Medical University (Other); Jiangxi Maternal and Child Health Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Second Affiliated Hospital of Zhengzhou University (Other); Shanxi Provincial Maternity and Children's Hospital (Other); First Affiliated Hospital of Guangxi Medical University (Other); Guangxi Maternal and Child Health Hospital (Other); Yinchuan Municipal Maternal and Child Health Hospital (Unknown); Xinjiang Jiayin Hospital (Unknown)
Responsible Party: Principal Investigator, Jiang Li, attending doctor, Peking University People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: prolonged down regulation
Record Dates: First submitted 2019-01-15; First posted 2019-01-18 (Actual); Last update posted 2019-01-18 (Actual); Status verified 2019-01

CONDITIONS: Infertility, Female
Keywords: down-regulation; controlled ovarian hyperstimulation; IVF/ICSI
MeSH Terms: conditions — Infertility, Female | interventions — Triptorelin Pamoate; Luteinizing Hormone

STUDY DESIGN:
Intervention Model Description: After the evaluation, patients met the eligible criteria will be informed, sign the consent form and be included in this study. We will randomly assign women (1:1) to early follicular phase prolonged down-regulation group (intervention group) or luteal phase long down-regulation group (control group), using a central randomization system with block sizes of 4 to 6 (changing constantly) and setting hospital as a stratification factor.
Who Masked: Outcomes Assessor
Masking Description: The researchers (physicians, nurses and embryologists) and patients are not blinded due to the nature of both interventions while the data analysts are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- early follicular phase down-regulation (Experimental): Patients have a injection of 3.75mg long-acting Triptorelin acetate (Dipherelin®, IPSEN, France) on the 1st-4th day of menstrual cycle. If complete pituitary down-regulation is achieved after 28-42 days, exogenous gonadotropins will be given according to the participants' BMI. The physician will monitor the follicular growth and adjust the dose of exogenous gonadotropins accordingly. When the desired follicle size is reached, human chorionic gonadotropin will be administered. Oocyte retrieval will be performed 36-38 hours after pre-ovulatory hCG injection transvaginally under ultrasound monitoring. Oocyte retrieved will be cultured in vitro for 3-6h before being fertilized via IVF or ICSI. Two top-quality Day 3 cleavage embryos will be transferred 72h after retrieval.
  Interventions: Drug: Triptorelin acetate
- luteal phase down-regulation (Active Comparator): Patients have a injection 0.1mg short-acting Triptorelin acetate (Decapeptyl®, Ferring, Germany) every day, 10-12 days before the next menstrual cycle. If complete pituitary down-regulation is achieved after 14-21 days, exogenous gonadotropins will be given according to the participants' BMI. The physician will monitor the follicular growth and the serum hormone level and adjust the dose of exogenous gonadotropins accordingly. When the desired follicle size is reached, human chorionic gonadotropin will be administered. Oocyte retrieval will be performed 36-38 hours later under ultrasound monitoring. Oocyte retrieved will be cultured in vitro for 3-6h before being fertilized via IVF or ICSI. Two top-quality Day 3 cleavage embryos will be transferred 72h after retrieval.
  Interventions: Drug: Triptorelin acetate

INTERVENTIONS:
Drug: Triptorelin acetate — Achieve pituitary down regulation with triptorelin acetate and start controlled ovarian stimulation after complete pituitary down regulation
  Other Names: recombinant follicular stimulating hormone (rFSH); recombinant luteinizing hormone (rLH); urinanry human postmenopausal gonadotropin (HMG)

SUMMARY:
Since the first "tube baby", Louise Brown, was born in the United Kingdom in 1978, many infertile couples have been benefitted from in vitro fertilization and embryo transfer (IVF-ET) and intracytoplasmic sperm injection (ICSI). Although a late starter, China is developing rapidly in ART and playing a more and more important role in the area of reproductive medicine.

In spite of the continuous development in ART, so far, the overall success rate of IVF/ICSI is still hovering around 25-40%. There are many factors influencing the success rate of IVF/ICSI. Among them, an appropriate controlled ovarian hyperstimulation (COH) protocol is directly associated with the number of oocyte retrieved, as well as the number and quality of embryos, which exert an important influence on the success rate of IVF/ICSI. The luteal phase pituitary down-regulation protocol is one of the most widely used COH protocols in clinical practice, particularly in China. Though effective, it may lead to an increased incidence of ovarian hyperstimulation syndrome (OHSS), as well as a negative impact on endometrial receptivity. The coping strategy is to freeze all the embryos and transfer in the next cycle. Though avoiding the above mentioned adverse effects, such strategy increases the time to pregnancy (TTP) and therefore results in certain psychological and economic burdens for infertile couples.

In recent years, some Chinese researches applied the early follicular full-dose down-regulation protocol that is always performed to women with endometriosis to a more general IVF/ICSI population and found a clinical pregnancy rate of 64% in the fresh embryo transfer cycle, much higher than that of the luteal phase down-regulation protocol. Furthermore, since this protocol decrease the risk of progesterone elevation on hCG day, it increases the fresh embryo transfer rate and shortens TTP.

Given most studies regarding the effectiveness and safety of the early follicular phase full-dose down-regulation protocol are retrospective studies, the results may be biased by several confounding factors. Therefore, we would like to conduct a multicenter, randomized controlled trial to compare the pregnancy outcome and safety indicators between the early follicular phase full-dose down-regulation protocol and the luteal phase down-regulation protocol.

DETAILED DESCRIPTION:
Background:

Since the first "tube baby", Louise Brown, was born in the United Kingdom in 1978, many infertile couples have been benefitted from in vitro fertilization and embryo transfer (IVF-ET) and intracytoplasmic sperm injection (ICSI). It is reported that there are over 5 million babies born with the help of assisted reproductive technology (ART). According to the 2015 national data published by Human Fertility and Embryology Authority (HFEA, 48,147 women received 61,726 IVF/ICSI cycles and gave birth to 17,041 newborns. In the United States, 169,602 IVF/ICSI cycles were performed in 2014 and 68,791 tubal babies were born. China has a huge population base, and therefore has a substantial number of infertile couples. Although a late starter, China is developing rapidly in ART and playing a more and more important role in the area of reproductive medicine.

In spite of the continuous development in ART, so far, the overall success rate of IVF/ICSI is still hovering around 25-40%. The live birth rate per stimulated cycle is 25.6% in the UK in 2015, fluctuating from 1.9% in women aged 45 and elder to 32.2% in women younger than 35 years old. The IVF/ICSI success rate in 2014 in the US is similar. In China, according to the data submitted by 115 reproductive medicine centers on the ART data reporting system developed by Chinese Society of Reproductive Medicine, the delivery rate is about 40%. Hence, there is much room for improvement regarding the live birth rate of IVF/ICSI, which is of great significance to infertile couples.

There are many factors influencing the success rate of IVF/ICSI, e.g. the infertile couples' age, the controlled ovarian hyperstimulation (COH) protocol, the quality and number of embryos for transferring, the endometrium and luteal phase support protocol, etc.. Among them, an appropriate COH protocol is directly associated with the number of oocyte retrieved, as well as the number and quality of embryos, which exert an important influence on the success rate of IVF/ICSI. The luteal phase pituitary down-regulation protocol is one of the most widely used COH protocols in clinical practice, particularly in China. In this protocol, gonadotropin releasing hormone agonist (GnRHa) administered in the previous luteal phase induces a state of down regulation of the pituitary gland via competitive occupying and further exhausting the GnRH receptors in the pituitary, which inhibits the endogenous luteinizing hormone (LH) peak and avoid spontaneous ovulation, decreasing the cycle cancellation rate. But the classic down-regulation protocol may lead to an increased incidence of ovarian hyperstimulation syndrome (OHSS), as well as a negative impact on endometrial receptivity due to the progesterone elevation after multiple oocytes development. The coping strategy is to freeze all the embryos and transfer in the next cycle. Though avoiding the above mentioned adverse effects, such strategy increases the time to pregnancy (TTP) and therefore results in certain psychological and economic burdens for infertile couples.

In recent years, some Chinese researches applied the early follicular down-regulation protocol that is always performed to women with endometriosis to a more general IVF/ICSI population and found a clinical pregnancy rate of 64% in the fresh embryo transfer cycle, much higher than that of the luteal phase down-regulation protocol. The possible mechanism is that it may improve the down regulation of LH and the endometrial receptivity, therefore having a better control of LH during COH, increasing the endometrial thickness on hCG day, as well as the embryo implantation rate and clinical pregnancy rate. Furthermore, since this protocol decrease the risk of progesterone elevation on hCG day, it increases the fresh embryo transfer rate and shortens TTP.

Objective:

Given most studies regarding the effectiveness and safety of the early follicular phase down-regulation protocol are retrospective studies, the results may be biased by several confounding factors. Therefore, we would like to conduct a multicenter, randomized controlled trial to compare the pregnancy outcome and safety between the early follicular phase and luteal phase down-regulation protocols.

Study design:

1. Screening： 1) Evaluation: vital signs, physical examination, laboratory test (routine tests+ AMH+ chromosome) and ultrasound examination (evaluating the ovarian reserve function); 2) Screening: to decide whether the women can be included in the study or not; 3) Collection of basic information (via electronic medical records and questionnaires): demographic characteristics, the history of infertility, menstrual, marriage and childbearing, the past history and surgery history, and the history of adverse environmental exposure;
2. Inclusion and randomization: After the evaluation, patients met the eligible criteria will be informed, and those who sign the consent form will be included in this study. We will randomly assign women (1:1) to early follicular phase down-regulation group (intervention group) or luteal phase down-regulation group (control group), using a central randomization system with block sizes of 4 to 6 (changing constantly) and setting hospital as a stratification factor.
3. Blinding: The researchers (physicians, nurses and embryologists) and patients are not blinded due to the nature of both interventions while the data analysts are blinded.
4. Intervention and control: The treatment period is from the down-regulation day to the day of oocyte retrieval, and the participants receive one of the following treatments:

1) Early follicular phase prolonged down-regulation group (intervention group): Patients have a injection of 3.75mg long-acting GnRHa (Dipherelin®, IPSEN, France) on the 1st-4th day of menstrual cycle as pituitary down-regulation.

2) Luteal phase long down-regulation group (intervention group): Patients have a injection of short-acting GnRHa (Decapeptyl®, Ferring, Germany) 0.1mg per day, 10-12 days before the menstruation as pituitary down-regulation.

5. Embryo transfer and Luteal phase support: Patients will receive luteal phase support with intramuscular progesterone (60mg/day) since the day of oocyte retrieval. On day 3 after oocyte retrieval, two top quality cleavage-stage embryos will be transferred via a catheter under transabdominal ultrasound guidance. The patients will lie in bed for 15 minutes after the procedure. Luteal phase support will be switched to 8% progesterone sustained-releasing vaginal gel (Crinone®, Merck, Switzerland) 90mg and dydrogesterone (Duphaston®, AbbottBiologicals, Netherlands) 20mg per day and continued for at least 2 weeks. For those who get pregnancy, luteal phase support will be continued to 10 weeks of gestation. The dosage adjustment will be determined by physicians of each study site according to their personal experience.

6. Pregnancy evaluation and follow up: All the information will be recorded in our follow-up forms designed specifically for each follow-up visit.

1. Biochemical determination: 14±4 days after embryo transfer, serum β-hCG will be tested to determine pregnancy.
2. Clinical pregnancy determination: 28±4 days after embryo transfer, a transvaginal ultrasound scan will be performed to confirm the presence of fetal sac, yolk sac and fetal heart.
3. Ongoing pregnancy determination: A transvaginal ultrasound scan will be performed at 10-12 weeks of gestation to confirm ongoing pregnancy. The presence of first-trimester pregnancy complications (e.g. OHSS, ectopic pregnancy, miscarriage etc.) will be registered according to the participant's medical record and a telephone follow-up.
4. 28 weeks of gestation: A telephone follow-up will be conducted to collect the information regarding the second trimester pregnancy complications.
5. 37 weeks of gestation: A telephone follow-up will be conducted to collect the information regarding the third trimester pregnancy complications.
6. Delivery information: A telephone follow-up will be made to collect delivery information including gestational age, delivery mode, delivery complications and infant information such as birth weight, any birth defect, etc.
7. Postpartum information: Postpartum information includes complications of both the mother and the infant, which will be collected 6 weeks after delivery.

For those not receiving a fresh embryo transfer (e.g. due to OHSS), and those not achieving live birth and with surplus cryopreserved embryos, the outcome of frozen-thawed embryo transfer cycles will be followed up and recorded as well.

7. Outcome measures:

1) Main outcome: live birth rate (effective indicator) per stimulated cycle. 2) Secondary outcomes include effective and safety indicators. 8. Biostatistic analysis method and sample size calculation:

1. Sample size will be calculated based on superiority test: α=0.05, 1-β=0.80. The reported live birth rate is about 30%, while the live birth rate of the prolonged protocol is predicted to be around 40% based on previous retrospective studies. We set the delta value as 6%, and the ratio between groups will be 1:1; therefore, the sample size of each group is 851. Taking into consideration a drop rate of 10%, we expect to ultimately have a total of 1892 enrollees, with 946 participants in each group.
2. Statistical analysis method:

   1. Statistical description We will adopt descriptive statistical analysis to summarize the participants' demographic characteristics, physical examination, laboratory tests, other health information and the outcome indicators. The continuous variables will be described with means and standard deviation (or median and interquartile range), while the categorical variable will be described with frequency and percentage. The proportion of drop-off cases will be calculated and analyzed.
   2. Comparable analysis It will be used to compare the demographic and other baseline characteristics to make sure the comparability of the two groups. If the continuous variables follow the normal distribution, t test will be performed; if not, the rank sum test or a normal transformation will be performed. For the categorical variables, chi-square test or Fisher's exact test will be performed.
   3. Statistical analysis for the outcome measures Between-group differences for categorical and continuous outcome variables will be assessed by logistic regression and linear regression, respectively.
   4. Safety analysis Adverse events and reaction will be listed and analyzed using the chi-square test.
   5. The analysis for the primary outcome and important outcome measurements will be based on both the intention-to-treat analysis and per-protocol analysis. The results of these two analyses will be compared in the final analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged between 20 to 35 years old and with a history of infertility (fail to get pregnant after over one year's regular, unprotected sex), who receive IVF/ICSI for one of the following reasons:

   ① Tubal factor: e.g. peritubal adhesions, tubal obstruction, etc.. Patients with hydrosalpinx can be enrolled after salpingectomy or tubal ligation;

   ② Male factor: e.g. oligospermia, asthenozoospermia, teratozoospermia, etc.;

   ③ Unexplained infertility: patients with a history of infertility more than 1 year but with no specific cause for infertility (ovulation, tubal, endometrial and male factor), or still not get pregnant after the above-mentioned causes being removed.
2. Women with a normal ovarian reserve according to: ①basal steroid hormone on day 2-4 of menstrual cycle: basal FSH≤10mIU/ml, estradiol (E2) <50pg/ml;②1.5<anti-Müllerian hormone (AMH)<4.0；③8≤antral follicle count (AFC) ≤15;
3. First IVF/ICSI cycle;
4. BMI≥18 and ≤25kg/m2;
5. Informed consent

Exclusion Criteria:

1. Women with a negative reproductive history, including a history of:

   ① recurrent miscarriage: women with twice and more than twice spontaneous miscarriage, missed abortion, biochemical pregnancies, etc.;

   ② fetal malformation or chromosomal abnormalities;

   ③ intrauterine death.
2. Women with a history of one side adnexectomy;
3. Women with a poor ovarian response or diminished ovarian reserve (based on Bologna' criteria);
4. Women with ovulation dysfunction;
5. Women with PCOS (based on Rotterdam's criteria);
6. Women with endometriosis;
7. Women with the following uterine abnormalities: uterine malformation (unicornuate uterus, uterus bicornis, uterus duplex, mediastinum uterus), adenomyosis, submucosa myoma, intrauterine adhesion;
8. Chromosomal abnormality for either or both of the couple;
9. Women with contraindications for ART or pregnancy: uncontrolled diabetes mellitus, cardiac disease, undiagnosed liver and/or renal function, vaginal bleeding, suspected or a past history of cervical cancer, endometrial cancer, breast cancer, and a history of deep venous thrombosis, pulmonary embolism, stroke, etc.;
10. Women who are enrolled in other clinical trials.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1892 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2020-09-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
live birth rate per transferred cycle | 28 weeks of gestation
  the number of live births (after 28 gestational week) divided by the number of transferred fresh cycles ×100%;

SECONDARY OUTCOMES:
live birth rate per stimulated cycle | 28 gestational week
  the number of live births (after 28 gestational week) divided by the number of all patients who started COH×100%
biochemical pregnancy rate per stimulated cycle | 12-15 days after embryo transfer
  the number of patients with a serum beta hCG of at least 10mIU/ml divided by the number of all patients who started COH ×100%
clinical pregnancy rate per stimulated cycle | 28-30 days after embryo transfer
  the number of patients with a intrauterine gestational sac divided by the number of all patients who started COH×100%
ongoing pregnancy rate per stimulated cycle | 10-12 weeks of gestation
  the number of patients with a viable intrauterine pregnancy divided by the number of all patients who started COH×100%
biochemical pregnancy rate per transferred cycle | 12-15 days after embryo transfer
  the number of patients with a serum beta hCG of at least 10mIU/ml divided by the number of transferred fresh cycles ×100%
clinical pregnancy rate per transferred cycle | 28-30 days after embryo transfer
  the number of patients with a intrauterine gestational sac divided by the number of transferred cycles×100%
ongoing pregnancy rate per transferred cycle | 10-12 weeks of gestation
  the number of patients with a viable intrauterine pregnancy divided by the number of transferred fresh cycles×100%
pregnancy loss rate | till 28 weeks of gestation
  the number of miscarriage and intrauterine fetal death cases divided by the number of participants with clinical pregnancy

OTHER OUTCOMES:
the incidence of moderate to severe OHSS | since oocyte retrieval to 13 weeks gestation
  the number of severe OHSS cases divided by the number of participants receiving oocyte retrieval
pregnancy complications | since embryo transfer to delivery (during pregnancy)
  all the complications occurred during pregnancy, e.g. preeclampsia, gestational diabetes, etc.
adverse fetal outcomes | 1 month after delivery
  all the recorded adverse fetal outcomes, e.g. fetal malformation etc
neonatal birth weight | at delivery
  birth weigh of the neonate at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Huan Shen, MD,phD, Principal Investigator — Peking University; Li Jiang, MD,MPH, Principal Investigator — Peking University

REFERENCES:
- [Background] The United Kingdom national data. Human Fertility and Embryology Authority. 2015
- [Background] The United States national assisted reproductive technology(ART) data. Centers for Disease Control and Prevention.2015
- [Background] Chinese Reproductive Medicine Society national assisted reproductive technology (ART) data. 2015
- [Background] L Hu, Y Sun. The impact of various controlled ovarian hyperstimulation (COS) protocols on the outcome of in vitro fertilization and embryo transfer (IVF-ET). Journal of Practical Obstetrics and Gynecology. 2014;30(10);723-725.
- [Background] Y Hu, T Ding, Y Zhao, Q Wu. The comparison of the birth outcome of in vitro fertilization and embryo transfer (IVF-ET) after two different down-regulation protocols. Maternal and Child Health Care of China.2017;32(4):808-810.
- [Background] D Xu, Q Wu. The comparison of the application of ultra-long down-regulation protocol and antagonist protocol in in vitro fertilization and embryo transfer (IVF-ET). Jiangxi Medical Journal. 2015;50(1):13-15.
- [Background] Q Su, Q Wu, L Tian, Y Li. The clinical analysis of different controlled ovarian hyperstimulation (COS) protocols in in vitro fertilization and embryo transfer (IVF-ET). Jiangxi Medical Journal. 2014;49(8):723-725.
- [Background] Y Li, Q Wu, Y Yi. The impact of the follicular phase ultra-long long down-regulation protocol on PCOS patients' outcome after in vitro fertilization and embryo transfer (IVF-ET). Jiangxi Medical Journal. 2014;49(2):117-120.
- [Background] L Nie, Q Wu, Y Zhang, J Chen. The analysis of the application of the follicular phase ultra-long down-regulation protocol in patients with fine ovarian reserve but a failed previous in vitro fertilization (IVF)/ intracytoplasmic sperm injection (ICSI) and embryo transfer. Progress in Obstetrics and Gynecology. 2011;20(6):470-472.
- [Background] F Gong, K Luo, G Lu. The effectiveness of the modified ultra-long down-regulation protocol in PCOS patients receiving in vitro fertilization and embryo transfer (IVF-ET). Basic and Clinical Medicine. 2010，30(9)：984-987.
- [Background] Moher D, Hopewell S, Schulz KF, Montori V, Gotzsche PC, Devereaux PJ, Elbourne D, Egger M, Altman DG; Consolidated Standards of Reporting Trials Group. CONSORT 2010 Explanation and Elaboration: Updated guidelines for reporting parallel group randomised trials. J Clin Epidemiol. 2010 Aug;63(8):e1-37. doi: 10.1016/j.jclinepi.2010.03.004. Epub 2010 Mar 25. PMID 20346624

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT03809221/Prot_SAP_000.pdf